CLINICAL TRIAL: NCT07137377
Title: CESARCOM Study Protocol: Assessing the Impact of Therapeutic Communication on Patients' Anxiety During Elective Cesarean Sections, - a Before-and-after Interventional Study
Brief Title: Assessing the Impact of Therapeutic Communication on Patients' Anxiety During Elective Cesarean Sections
Acronym: CESARCOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Océane Pécheux, Principal investigator, University Hospital, Geneva
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: ID 2024-02495; PRD 05-2024-II (Other Grant/Funding Number: Research and development Fund - University Hospitals of Geneva)
Record Dates: First submitted 2025-08-12; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Communication; Anxiety
Keywords: hypnosis based therapeutic communication; anxiety; STAI score
MeSH Terms: conditions — Communication; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients' anxiety before and after a teaching programme of the providers.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients' do not know if they are in the pre intervention group or in the post intervention group. The statistician will not know which is the pre or the post intervention group either.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre intervention group (before hypnosis-based therapeutic communication reaching programme) (No Intervention): Patients' anxiety levels before the implementation of an online teaching programme about hypnosis based therapeutic communication in obstetrics.
- post intervention group (after hypnosis-based therapeutic communication teaching programme) (Experimental): Patients' anxiety levels after the implementation of an online teaching programme about hypnosis based therapeutic communication in obstetrics.
  Interventions: Behavioral: On line teaching CESARCOM teaching programe (immersive podcasts, digital flashcards)

INTERVENTIONS:
Behavioral: On line teaching CESARCOM teaching programe (immersive podcasts, digital flashcards) — A short e-learning program (immersive podcasts, digital flashcards) will be carried out for the medical and paramedical staff of the cesarean section operating room, by a specialized team. It will will consist of :
  * the presentation of the basic principles of therapeutic communication (listening, empathy, verbal, non-verbal, paraverbal language)
  * the distribution of the "HUG communication lexicon/wordbook" .
  * educational scenes illustrating the impact of therapeutic communication in the operating room ("good" versus "bad" words).
  Arms: post intervention group (after hypnosis-based therapeutic communication teaching programme)

SUMMARY:
Background:

Anxiety is highly prevalent before elective caesarean sections and can have a negative impact on anesthetic outcomes, postoperative pain and maternal mental health. The use of pharmacological premedication is controversial, and non-pharmacological alternatives are increasingly being explored. Therapeutic communication, based on empathy, positive language and the conscious avoidance of negative or anxiety-inducing suggestions, has shown promise in other surgical settings. However, its effectiveness in obstetrics remains to be explored.

Methods This is a single-centre, prospective, observational, before-and-after study. The study aims to assess whether implementing an on-line (asynchronous) training programme on therapeutic communication for obstetric care teams can reduce maternal anxiety following elective caesarean sections. The study includes two groups of 130 patients each, one before the intervention and one after. Anxiety levels will be assessed using the French version of the State-Trait Anxiety Inventory score, and the primary outcome will be the difference in scores after caesarean section between the two groups. Secondary outcomes include the proportion of patients with high anxiety levels (STAI-State score >45), as well as staff satisfaction, feeling of relevance, and indicators of the feasibility of implementing the training.

The intervention consists of a short (less than 1 hour) training course using podcasts and flashcards, combined with distributing a lexicon that promotes hypnosis-based therapeutic communication (HBTC). Staff participation, perceived relevance and satisfaction will be assessed using structured questionnaires based on the Likert scale.

Linear and logistic regression analyses will be used to adjust for confounding variables, including baseline anxiety, psychiatric history, and intraoperative complications.

Discussion This is the first study to evaluate the impact of a dedicated HBTC training programme on patient anxiety and staff experience in an obstetric surgical setting. By integrating this approach into routine cesarean section care, our aim is to improve the patient experience and enhance communication practices within clinical teams. The results could inform clinical practices on non-pharmacological strategies in obstetric care.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years

* elective c-section planned in the Maternity Unit of the Geneva University Hospitals
* consent to participate

Exclusion Criteria:

* Not-French-speaking patients (interpreter required).
* All emergency c-sections.
* Death during the intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Post elective cesarean anxiety level | Within 24 hours after cesarean.
  To assess the impact of a therapeutic communication wordbook and hypnosis-based therapeutic communication teaching programme on patients' anxiety levels after elective c-section and the proportion of elevated anxiety levels after elective c-sections, before and after implementation of a therapeutic communication protocol/short teaching programme.
  Patients' will receive State-State Anxiety Inventory (STAI) scores by email and complete them on line. Their result will be directly transfer to REDCap, data management software.
  We will report difference of means of the post c-section anxiety assessed with the STAI score (as a continuous variable), each patient result being adjusted on its pre c-section STAI score (result at baseline).
  Minimum STAI score result=20; maximum=80. The higher the score, the greater the level of anxiety.

SECONDARY OUTCOMES:
High anxiety levels proportion | Within the 24 hours after cesareans.
  Differences of proportions of patients with a post- c-section State Anxiety Inventory (STAI-S) score > 45 in the two groups, and to assess the providers satisfaction with the teaching programme, as long as the feasibility of implementing such a programme in obstetrics.
Providers satisfaction | At 6 and 12 months after the programme
  The satisfaction of the team (comprising nurses, midwives, doctors, and residents) will be measured using Likert scales (minimum result=10; maximum=50; the higher is the score, the greater the level of satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- HUG, Geneva, Switzerland

REFERENCES:
- [Background] Gaudry E, Vagg P, Spielberger CD. Validation of the State-Trait Distinction in Anxiety Research. Multivariate Behav Res. 1975 Jul 1;10(3):331-41. doi: 10.1207/s15327906mbr1003_6. PMID 26829634
- [Background] Lang EV, Hatsiopoulou O, Koch T, Berbaum K, Lutgendorf S, Kettenmann E, Logan H, Kaptchuk TJ. Can words hurt? Patient-provider interactions during invasive procedures. Pain. 2005 Mar;114(1-2):303-9. doi: 10.1016/j.pain.2004.12.028. Epub 2005 Jan 26. PMID 15733657
- [Background] Caddick J, Jawad S, Southern S, Majumder S. The power of words: sources of anxiety in patients undergoing local anaesthetic plastic surgery. Ann R Coll Surg Engl. 2012 Mar;94(2):94-8. doi: 10.1308/003588412X13171221501267. PMID 22391371
- [Background] Varga K. Suggestive techniques connected to medical interventions. Interv Med Appl Sci. 2013 Sep;5(3):95-100. doi: 10.1556/IMAS.5.2013.3.1. Epub 2013 Sep 16. PMID 24265898
- [Background] Boselli E, Demaille N, Fuchs G, Manseur A. [Assessment of the therapeutic communication in order to improve the welcoming of patients in the operating room: impact study]. Can J Anaesth. 2018 Oct;65(10):1138-1146. doi: 10.1007/s12630-018-1167-2. Epub 2018 Jun 11. French. PMID 29949092
- [Background] Wilson CJ, Mitchelson AJ, Tzeng TH, El-Othmani MM, Saleh J, Vasdev S, LaMontagne HJ, Saleh KJ. Caring for the surgically anxious patient: a review of the interventions and a guide to optimizing surgical outcomes. Am J Surg. 2016 Jul;212(1):151-9. doi: 10.1016/j.amjsurg.2015.03.023. Epub 2015 Jun 2. PMID 26138522
- [Background] Hishikawa K, Kusaka T, Fukuda T, Kohata Y, Inoue H. Anxiety or Nervousness Disturbs the Progress of Birth Based on Human Behavioral Evolutionary Biology. J Perinat Educ. 2019 Oct 1;28(4):218-223. doi: 10.1891/1058-1243.28.4.218. PMID 31728113
- [Background] Kassahun WT, Mehdorn M, Wagner TC, Babel J, Danker H, Gockel I. The effect of preoperative patient-reported anxiety on morbidity and mortality outcomes in patients undergoing major general surgery. Sci Rep. 2022 Apr 15;12(1):6312. doi: 10.1038/s41598-022-10302-z. PMID 35428818
- [Background] Schaal NK, Fehm T, Wolf OT, Gielen P, Hagenbeck C, Heil M, Fleisch M, Hepp P. Comparing the course of anxiety in women receiving their first or repeated caesarean section: A prospective cohort study. Women Birth. 2020 May;33(3):280-285. doi: 10.1016/j.wombi.2019.05.011. Epub 2019 Jun 6. PMID 31176587
- [Derived] Pecheux O, Vocat M, Coen M, de Oliveira S, Bouscail Hardy AL, Jaksic C, Silvestrini N, Campelo S, Othenin-Girard V, Montandon-La-Longe CY, Chilin A, Suppan M, Al Khoury Al Kallab R, Daelemans C. CESARCOM study protocol: assessing the impact of therapeutic communication on patients' anxiety during elective cesarean sections, - a before-and-after interventional study. BMC Pregnancy Childbirth. 2025 Oct 14;25(1):1082. doi: 10.1186/s12884-025-08193-9. PMID 41088028